CLINICAL TRIAL: NCT04271748
Title: The Impact of Time Restricted Feeding in Crohn's Disease
Acronym: TRF-CD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: The Kenneth Rainin Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-11021081
Record Dates: First submitted 2020-02-13; First posted 2020-02-17 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Crohn's Disease (CD)
Keywords: Fasting; Time Restricted Feeding; Intermittent Fasting; Inflammatory Bowel Diseases (IBD); IBD; CD
MeSH Terms: conditions — Crohn Disease; Fasting; Intermittent Fasting; Inflammatory Bowel Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Time Restricted Feeding (Experimental): Subjects will be required to fast for 16 consecutive hours daily for 4 weeks. The registered dietitian will provide subjects counseling on the intermittent fasting regimen.
  Interventions: Other: Time Restricted Feeding

INTERVENTIONS:
Other: Time Restricted Feeding — The counseling on the regimen will involve instructing the subjects on study compliance and fasting times. Subjects will be instructed to choose an eight-hour eating window (e.g., 11:00am - 7:00pm) during which the patient will be able to eat his/her normal diet. During the 16-hour fasting window (e.g., 7:00pm - 11:00am), the participant will be able to drink regular water and black coffee.
  Other Names: Intermittent Fasting

SUMMARY:
Time-restricted feeding (TRF) is a dietary regimen involving the consumption of food and liquids within a defined time window with or without additional restriction on dietary composition. TRF has been associated with improvements in inflammation, host metabolism, autophagy, gut microbial composition, and gut permeability. Crohn's disease is an inflammatory bowel disease of unknown etiology that likely results from a combination of genetic and environmental factors. This proposed study will test the hypothesis that a time-restricted feeding regimen will improve clinical outcomes and favorably influence the gut microbiome in patients with active Crohn's disease. If time-restricted fasting proves beneficial to this patient population then it will pave the way for larger, prospective studies and clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Subjects has active Crohn's disease of the ileum and/or colon. The diagnosis should be confirmed by endoscopic or radiological evidence.
* Active inflammation on colonoscopy performed as evidenced by an SES-CD ≥ 6 (or ≥ 4 for isolated ileal disease) OR C-Reactive protein ≥ 1.0 mg/L OR fecal calprotectin ≥ 250 μg/g. Any or all of these results must be from within 180 days of study entrance.
* Subject should have BMI of >18.5 and <40

Exclusion Criteria:

* Subjects who decline to provide informed consent
* Subject with a history of an eating disorder, major gastrointestinal surgery within the past 3 months.
* Subject with a history of antibiotic use within 4 weeks.
* Subject with a history of bowel obstruction within the past 12 months
* Subject with a history of diabetes requiring medication
* Subject who is currently pregnant or breastfeeding will be excluded
* Subjects with current antibiotic use. In order to participate, subjects will be required to have a 2-week wash-out period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-01-14 (Actual); Primary Completion 2022-08-16 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Change in patient reported outcomes as measured by Patient Recorded Outcome 2 (PRO2) scores. | Baseline (Week 0); 4 weeks after incorporating time restricted feeding into diet
  This will be measured to assess clinical response as determined by a reduction of either 8 or more points or a total PRO2 score of less than or equal to 8 points. The PRO2 score scale ranges from a score of 0 as the minimum and has no maximum limit. A score below 8 is considered remission; a score less than 14 is considered mild; and a score greater than 34 is considered severe.
Change in Inflammatory Markers as measured by blood C-reactive protein (CRP). | Baseline (Week 0); 4 weeks after incorporating time restricted feeding into diet
  This will be measured to assess clinical response as determined by a reduction of 50% or more from baseline or normalization of the CRP level results.
Change in inflammatory markers as measured by fecal calprotectin lab results | Baseline (Week 0); 4 weeks after incorporating time restricted feeding into diet
  This will be measured to assess clinical changes as determined by a reduction of 50% or more from baseline or normalization of the calprotectin levels results.

SECONDARY OUTCOMES:
Change in taxonomic composition of the gut microbiome as measured by Polymerase Chain Reaction (PCR) analysis. | Baseline (Week 0); 4 weeks after incorporating time restricted feeding into diet
  This will be measured to assess the impact of time restricted feeding on intestinal microbiota composition.
Markers of systemic peripheral blood immunity as measured by Mass Cytometry by Time-Of-Flight (CyTOF) analysis. | Baseline (Week 0); 4 weeks after incorporating time restricted feeding into diet
  This will be measured to assess the effect of time restricted feeding on immune cell composition.

CONTACTS AND LOCATIONS:
Overall Officials: Dana J Lukin, MD, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Celiberto LS, Graef FA, Healey GR, Bosman ES, Jacobson K, Sly LM, Vallance BA. Inflammatory bowel disease and immunonutrition: novel therapeutic approaches through modulation of diet and the gut microbiome. Immunology. 2018 Sep;155(1):36-52. doi: 10.1111/imm.12939. Epub 2018 May 16. PMID 29693729
- [Background] Mattson MP, Longo VD, Harvie M. Impact of intermittent fasting on health and disease processes. Ageing Res Rev. 2017 Oct;39:46-58. doi: 10.1016/j.arr.2016.10.005. Epub 2016 Oct 31. PMID 27810402
- [Background] Patterson RE, Sears DD. Metabolic Effects of Intermittent Fasting. Annu Rev Nutr. 2017 Aug 21;37:371-393. doi: 10.1146/annurev-nutr-071816-064634. Epub 2017 Jul 17. PMID 28715993
- [Background] Nagai M, Noguchi R, Takahashi D, Morikawa T, Koshida K, Komiyama S, Ishihara N, Yamada T, Kawamura YI, Muroi K, Hattori K, Kobayashi N, Fujimura Y, Hirota M, Matsumoto R, Aoki R, Tamura-Nakano M, Sugiyama M, Katakai T, Sato S, Takubo K, Dohi T, Hase K. Fasting-Refeeding Impacts Immune Cell Dynamics and Mucosal Immune Responses. Cell. 2019 Aug 22;178(5):1072-1087.e14. doi: 10.1016/j.cell.2019.07.047. PMID 31442401
- [Background] Jordan S, Tung N, Casanova-Acebes M, Chang C, Cantoni C, Zhang D, Wirtz TH, Naik S, Rose SA, Brocker CN, Gainullina A, Hornburg D, Horng S, Maier BB, Cravedi P, LeRoith D, Gonzalez FJ, Meissner F, Ochando J, Rahman A, Chipuk JE, Artyomov MN, Frenette PS, Piccio L, Berres ML, Gallagher EJ, Merad M. Dietary Intake Regulates the Circulating Inflammatory Monocyte Pool. Cell. 2019 Aug 22;178(5):1102-1114.e17. doi: 10.1016/j.cell.2019.07.050. PMID 31442403
- [Background] MacLellan A, Moore-Connors J, Grant S, Cahill L, Langille MGI, Van Limbergen J. The Impact of Exclusive Enteral Nutrition (EEN) on the Gut Microbiome in Crohn's Disease: A Review. Nutrients. 2017 May 1;9(5):447. doi: 10.3390/nu9050447. PMID 28468301
- [Background] Suskind DL, Cohen SA, Brittnacher MJ, Wahbeh G, Lee D, Shaffer ML, Braly K, Hayden HS, Klein J, Gold B, Giefer M, Stallworth A, Miller SI. Clinical and Fecal Microbial Changes With Diet Therapy in Active Inflammatory Bowel Disease. J Clin Gastroenterol. 2018 Feb;52(2):155-163. doi: 10.1097/MCG.0000000000000772. PMID 28030510
- [Background] Khanna R, Zou G, D'Haens G, Feagan BG, Sandborn WJ, Vandervoort MK, Rolleri RL, Bortey E, Paterson C, Forbes WP, Levesque BG. A retrospective analysis: the development of patient reported outcome measures for the assessment of Crohn's disease activity. Aliment Pharmacol Ther. 2015 Jan;41(1):77-86. doi: 10.1111/apt.13001. Epub 2014 Oct 27. PMID 25348809